CLINICAL TRIAL: NCT00276315
Title: A Phase III, Multicentre, Randomised, Assessor-blind, Parallel Groups, Reference Drug Controlled Study to Assess the Efficacy and Safety of a Single Administration, by Subcutaneous Injection of Dysport® for the Treatment of Hemifacial Spasm
Brief Title: Assessment of Effectiveness and Safety of Dysport® for the Treatment of Hemifacial Spasm
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-38-52120-074
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Hemifacial Spasm
MeSH Terms: conditions — Hemifacial Spasm | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

INTERVENTIONS:
Biological: Botulinum toxin type A
  Other Names: AbobotulinumtoxinA (Dysport®)

SUMMARY:
To compare the effectiveness and safety of Dysport® with the domestic Botulinum Toxin Type A (manufactured by Lanzhou Biologic Product Institute, P.R. China) for the treatment of hemifacial spasm.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from hemifacial spasm with at least 6 months duration (prior to visit 1)
* Cohen scale ≥ to grade II

Exclusion Criteria:

* Botulinum toxin type A treatment history within last 16 weeks prior to visit 1
* Hemifacial spasm secondary to facial palsy
* Previous alcohol or phenol injections or surgical therapy of the facial muscles
* Requirement for botulinum toxin injection to site(s) of the body other than in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2005-12; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Percentage of responders (defined as Cohen scale improvement ≥ to 2 levels) | At the end of week 4

SECONDARY OUTCOMES:
Percentage of responders (defined as Cohen scale improvement ≥ to 2 levels after medication) | At the end of week 1 and 12
Improvement degree of spasm (Jankovic scale) | At the end of week 1, 4 and 12
Assessment of efficacy by the subjects | At the end of week 1, 4 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (4):
- China (4):
  - Neurology Department, Peking Union Medical College Hospital, Beijing
  - Neurology Department, Guangdong Provincial People's Hospital, Guangdong
  - Neurology Department, Sir Run Run Shaw Hospital, Zhejiang University, Hangzhou
  - Neurology Department, Shanghai Ruijin Hospital, Shanghai